CLINICAL TRIAL: NCT05293990
Title: Usefulness of Gadovist-enhanced FLAIR Imaging in Differentiation Between a Glioblastoma and Solitary Brain Metastasis: Single Center Prospective Study
Brief Title: Usefulness of Gadovist-enhanced FLAIR Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryoo, In Seon (Other)
Responsible Party: Sponsor-Investigator, Ryoo, In Seon, Associate Professor of Radiology, Korea University Guro Hospital
Organization: Korea University Guro Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017GR0776
Record Dates: First submitted 2022-02-08; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Malignant Tumors; Brain Lymphoma; CNS Lymphoma
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: For a single malignant mass in the brain, conventional T1 highlighted contrast enhancement findings and histological results (glioblastoma/metastatic brain cancer) were compared and analyzed, followed by diagnosing a single brain mass (Df/Dt1, Dt2/Dt1, Dt2/Df ratio) and histological results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast-enhanced fluid attenuated inversion recovery (Other): Confirmation of the difference between FLAIR contrast enhancement and T1 contrast enhancement patterns-->PACS monitor shows the maximum dimension of FLAIR and T1 contrast enhancement by two neurology radiologists on FLAIR and T1 contrast enhancement images. In addition, the maximum diameter of the T2 high-signal lesion around the tumor is obtained using FLAIR images before contrast in the same plane. (Dt2)
  Interventions: Radiation: Usefulness of Gadovist-enhanced FLAIR imaging in differentiation between a glioblastoma and solitary brain metastasis

INTERVENTIONS:
Radiation: Usefulness of Gadovist-enhanced FLAIR imaging in differentiation between a glioblastoma and solitary brain metastasis — Usefulness of Gadovist-enhanced FLAIR imaging in differentiation between a glioblastoma and solitary brain metastasis

SUMMARY:
Polyplastic glioblastoma and metastatic brain cancer are the most common malignant brain tumors in adults. The primary diagnostic test for tumors in the brain shows magnetic resonance imaging or similar imaging findings (especially single metastatic brain cancer) that make it difficult to distinguish between these two diseases. In addition, due to the specificity of the tissue called the brain, biopsy is not easy and sometimes biopsy is difficult, so non-invasive discrimination is often important, and it is important how much prediction is made before the biopsy. To solve this problem, various advanced magnetic resonance imaging techniques have been studied, but they are all tests that need to be additionally conducted on ordinary magnetic resonance images, and there are many subjective factors, so complex data and statistical processing methods, and many cannot be easily tested. In addition, in all of these tests, accuracy is still reported at around 60%. Therefore, if contrast-enhanced FLAIR images can be obtained along with contrast-enhanced T1 images performed during conventional magnetic resonance imaging tests to help differentiate between two diseases, it will greatly help diagnose and treat brain tumor patients and facilitate clinical application.

DETAILED DESCRIPTION:
Polyplastic glioblastoma and metastatic brain tumors are the most common brain tumors in adults. Polyplastic glioblastoma is the most common tumor among malignant primary brain tumors, and metastatic brain tumors are the most common brain tumors in adults. In the diagnosis of brain tumors, magnetic resonance imaging is the most basic and primary imaging technique to date. However, in the case of a single metastatic brain tumor, the tumor shape, signal intensity, contrast enhancement pattern, and peripheral signal intensity appear so similar that they are hardly distinguished from polymorphic glioblastoma in conventional magnetic resonance images. However, it is very important to distinguish between the two diseases because the above two diseases have completely different characteristics in clinical aspects, surgical method decisions, treatment decisions, and prognosis. Obtaining histological results will be the ultimate answer, but due to the nature of tissue called the brain, non-invasive tests are preferred, and sometimes patients (e.g., cardiovascular disease) or lesions themselves cannot handle surgery are in a very important part of the brain, so it depends on imaging techniques. In addition, the distinction between the two diseases through imaging is important in that it is important to predict in advance even if biopsy is performed through surgery. Therefore, various advanced magnetic resonance imaging techniques such as diffusion-enhanced imaging (DWI), perfusion imaging (perfusion), and spectroscopic imaging (MR spectroscopy) have been attempted to better differentiate the two diseases through imaging tests. However, these images are additional imaging tests that need to be obtained after obtaining conventional magnetic resonance images and are usually accompanied by complex and various statistical analyses due to many subjective elements. In addition, there are tests that are difficult to conduct other than large hospitals with a certain size or larger. Nevertheless, the accuracy of the discrimination between the two diseases to date is around 60%. In addition, such tests are often difficult to perform in most hospitals, except for large hospitals with a certain size or larger. Therefore, if the two diseases can be better identified in conventional magnetic resonance imaging, it will be of great help to patient care clinically and it is expected that actual clinical application will be easier. Contrast-enhanced T1 highlighted images are always performed in conventional magnetic resonance images, and after that, one more FLAIR image is obtained to see if contrast-enhanced FLAIR images are helpful in differentiating the two diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo treatment, including surgery, after examining contrast-enhanced MR with an intra-brain mass that must exclude malignant tumors.
* Adults over 19 years of age at the time of examination
* Patients who agreed to this clinical study

Exclusion Criteria:

* In the case of severe cognitive of dysfunction or neurological defects (mRS>3)
* Pregnant or lactating patient
* Patients who are allergic to MRI contrast agents or cannot perform MRI for other reasons.
* Patients participating in other drug clinical trials as of the screening day (observation studies are possible)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by axial FLAIR and axial spin-echo T1-weighted image | about 5 year
  Two 3.0 Tesla MR machines (MAGNETOM Trio A Tim and MAGNETOM Prisma; Siemens, Erlangen, Germany) were used in this study. The protocol consisted of axial FLAIR (TR/TE/TI=9,000/100/2,500 milliseconds, with slice thickness of 2 mm) and axial spin-echo T1-weighted image (TR/TE=675/8.9 milliseconds, with slice thickness of 2 mm). After both pre-enhancement images are acquired, CE-T1WI and CE-FLAIR sequences were obtained 5 and 10 minutes after administering gadolinium-based contrast agents, respectively. Gadobutrol (Gadovist™, 0.1 millimol per kilogram of body weight, Schering AG, Berlin, Germany) was used as the contrast agent, via automated injector (Spectris MR; Medrad Europe, Maastricht, Netherlands). Subtraction images for both CE-FLAIR and CE-T1WI sequences were also obtained. Detailed protocol image sequence parameter is provided in shown in Online Resource 2.

CONTACTS AND LOCATIONS:
Overall Officials: Ryoo In Seon, dotorate, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, Gurogu, South Korea